CLINICAL TRIAL: NCT04432844
Title: Ultrasound Guided Internal Jugular Vein Cannulation Using Biplanar Imaging: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Other Study IDs: IJV Protocol V2
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biplanar Ultrasound guided Internal Jugular Vein Cannulation — Using Philips EPIQ elite ultrasound system with a high-frequency 3D and 4D volume linear array transducer (USG XL 14-3) to obtain the biplanar imaging of Internal jugular vein cannulation.

SUMMARY:
Central Venous access by real-time ultrasound guidance is considered as gold standard and a recommended clinical practice. Internal jugular vein cannulation is one of the central venous access commonly used for major cardiac surgeries for monitoring and administering life-saving medications. In daily practice internal jugular vein cannulation is done under the guidance of ultrasound imaging after general anesthesia before the surgery. Real time 2D ultrasound guidance (USG) during central venous cannulation (CVC) has shown to be superior to the traditional anatomical landmark guided CVC, but the incidence of carotid puncture is still 4.2%. Any improvement that aids in the ease and safety of the procedures needs to be evaluated. Recently USG biplanar imaging can now successfully demonstrate real time imaging in two different views at the same time. Theoretically, this may help improve precision by improving real time needle tip visualization and thereby reduce potential complications as compared to a traditional 2D approach. This study aims to assess the feasibility of biplanar USG internal jugular venous cannulation.

DETAILED DESCRIPTION:
This is a single arm prospective observational pilot study conducted at Prince of Wales Hospital in Hong Kong SAR. 20 adult patients scheduled for elective cardiac surgeries under general anesthesia (GA) will be recruited. After GA, patients will be positioned in the head low position for the USG guided IJV access. The skin of the neck will be prepared in a standard aseptic fashion. After sterilization, the surrounding area will be covered with a full-body sterile drape. The footprint and the cable of the ultrasound transducer will also be covered with a sterile transparent cover. Sterile ultrasound gel will be used for acoustic coupling during the USG guided CVC placement, but care will be taken to avoid inserting the needle through the US gel.

USG XL 14-3 transducer will be used to obtain the biplanar imaging of IJV. A 3 lumen CVC will be used to access the IJV. An experienced anesthesiologist shall perform the USG guided procedure using the Seldinger method. This special transducer can provide real-time short axis (out of the plane) and long axis (In-plane) view which can be used to identify, locate and choose the introducer needle entry site for IJV vascular access. IJV will be assessed for any anatomical variations, pre-existing pathologies and patency. Among the 'out of plane' and 'in plane' view, the former will be used as a primary view to guide the CVC introducer needle. The reference mark/line in the primary 'out of the plane' image in the biplanar view can be adjusted sidewise to visualise the needle in the 'in plane' view. As the needle is visualised in the 'in plane' technique (figure 1), the relative position of the needle to the target IJV can be determined which will further help in redirecting the needle towards the IJV. Needle tip can be made visualised in the 'out of the plane' view by carefully moving the transducer initially towards the introducer needle. Once the needle tip is visualised, it is advanced further towards the target taking into consideration both the 'in plane' and 'out of plane' image guidance. When the needle is visualised (in both the views) inside the vein, the transducer will be kept aside, a 5 ml syringe will be used to aspirate blood and then the guidewire is inserted into the IJV. Presence of guidewire will be again confirmed using the same biplanar transducer before performing the dilatation of IJV and final passage of the CVC. Likewise, the final position of the CVC shall also be confirmed using biplanar imaging. After final confirmation, CVC will be secured safely to the neck using sutures and connected to the pressure transducers for central venous pressure (CVP) monitoring.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to III
* Patients posted for elective cardiac surgeries under general anaesthesia.

Exclusion Criteria:

* Patient refusal
* skin entry site infection
* history of previous IJV cannulation
* obese patients (BMI>30)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for elective cardiac surgeries that meet the inclusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Time taken for successful IJV cannulation | Procedure (before surgery after general anesthesia)
  The time taken from the skin puncture to the aspiration of blood

SECONDARY OUTCOMES:
number of skin puncture | from the start of IJV insertion till the end of the procedure
  the number of skin puncture for the procedure
number of needle re-directions | Procedure during IJV insertion
  changes in the direction of needle insertion without removing it from the skin

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hosptial, Shatin, New Territories, Hong Kong